CLINICAL TRIAL: NCT00914524
Title: An Open-label Study of Olmesartan Medoxomil (CS-866) in Normotensive Patients With Chronic Glomerulonephritis or Diabetic Nephropathy
Brief Title: Study of Olmesartan Medoxomil (CS-866) in Patients With Chronic Glomerulonephritis or Diabetic Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Yasuhiro Tomono, Daiichi Sankyo Co., Ltd.
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS0866-C-J201
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Glomerulonephritis; Diabetic Nephropathy
Keywords: Chronic Glomerulonephritis; Diabetic Nephropathy; Angiotensin II Receptor Blocker; Urinary Protein
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Olmesartan Medoxomil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): 16 weeks of treatment starting with 5 mg of olmesartan medoxomil. If tolerated, the dose was increased to the next higher dose at weeks 4, 8, and 12.
  Interventions: Drug: olmesartan medoxomil

INTERVENTIONS:
Drug: olmesartan medoxomil — olmesartan medoxomil tablets, once daily

SUMMARY:
The treatment period was 16 weeks, the initial dose, 5 mg, was unforcedly titrated to 10 mg, 20 mg and 40 mg after confirming tolerance at weeks 4, 8 and 12. The primary endpoint for efficacy was the change in the urinary protein/creatinine ratio from baseline to the end of treatment. The secondary endpoint was creatinine clearance (Ccr).

ELIGIBILITY:
Inclusion Criteria:

* urinary protein/creatinine ratio in the 0.50 g/g to 3.50 g/g creatinine range
* normal sitting blood pressure values: systolic blood pressure of 100 mmHg or above but below 140 mmHg; diastolic blood pressure of 50 mmHg or above but less than 90 mmHg

Exclusion Criteria:

* treatment with corticosteroids or immunosuppressants
* treatment with antihypertensives (other than ARBs and ACE inhibitors)
* serum potassium level of 5.5 mEq/l or above
* serum creatinine level of 2.0 mg/dl or above

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-01; Primary Completion 2006-04 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
The change in the urinary protein/creatinine ratio from baseline to the end of treatment. | baseline to 16 weeks

SECONDARY OUTCOMES:
The change of creatinine clearance | baseline to 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan